CLINICAL TRIAL: NCT01316237
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled, Multiple Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GS-6620 in Treatment Naïve Subjects With Chronic Hepatitis C Virus Infection
Brief Title: A Study Evaluating the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GS-6620 in Treatment Naïve Subjects With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-119-0101
Record Dates: First submitted 2011-02-03; First posted 2011-03-16 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; HCV RNA; Polymerase inhibitor; Treatment naïve; GS-6620
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — GS-6620; BID protein, human

ARMS (9):
- Cohort 1 (Other): (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2) 50 mg GS-6620 or placebo QD in the morning with food [total daily dose (TDD) = 50 mg] for 5 days
  Interventions: Drug: GS-6620
- Cohort 2 (Other): (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  100 mg GS-6620 or placebo QD in the morning with food (TDD = 100 mg) for 5 days
  Interventions: Drug: GS-6620
- Cohort 3 (Other): Cohort 3 (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  300 mg GS 6620 or placebo QD in the morning with food (TDD = 300 mg) for 5 days
  Interventions: Drug: GS-6620
- Cohort 4 (Other): Cohort 4 (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  100 mg GS 6620 or placebo QD in the morning without food (TDD = 100 mg) for 5 days
  Interventions: Drug: GS-6620
- Cohort 5 (Other): Cohort 5 (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  300 mg GS 6620 or placebo QD in the morning without food (TDD = 300 mg) for 5 days
  Interventions: Drug: GS-6620
- Cohort 6 (Other): Cohort 6 (N = 10, genotype 2 or genotype 3): (Active drug: 8, Matching Placebo: 2)
  900 mg GS 6620 or placebo QD in the morning without food (TDD = 900 mg) for 5 days
  Interventions: Drug: GS-6620
- Cohort 7 (Other): Cohort 7 (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  450 mg GS 6620 or placebo, administered BID with food (TDD = 900 mg) for 5 days
  Interventions: Drug: GS-6620 tablet, 450 mg BID
- Cohort 9 (Other): Cohort 9 (N = 10, genotype 1): (Active drug: 8, Matching Placebo: 2)
  900 mg GS 6620 or placebo BID in the with food (TDD = 1800 mg) for 5 days
  Interventions: Drug: GS-6620 tablet
- Cohort 11 (Other): Cohort 11 (N = 10, genotype 1 : (Active drug: 8, Matching Placebo: 2)
  Up to 450 mg GS-6620 or placebo as an oral solution, BID, 12 hours apart in the fasted state, 2 hours after a meal (up to TDD = up to 900 mg) for 5 days.
  Interventions: Drug: GS-6620 tablet

INTERVENTIONS:
Drug: GS-6620 — GS-6620 tablet, 50 mg QD
  Arms: Cohort 1
Drug: GS-6620 — GS-6620 tablet, 100 mg QD
  Arms: Cohort 2
Drug: GS-6620 — GS-6620 tablet, 300 mg QD
  Arms: Cohort 3
Drug: GS-6620 — GS-6620 tablet, 100 mg QD, Fasted
  Arms: Cohort 4
Drug: GS-6620 — GS-6620 tablet, 300 mg QD, Fasted
  Arms: Cohort 5
Drug: GS-6620 — GS-6620 tablet, 900 mg QD, Fasted
  Arms: Cohort 6
Drug: GS-6620 tablet, 450 mg BID — GS-6620 tablet, 450 mg BID
  Arms: Cohort 7
Drug: GS-6620 tablet — GS-6620 tablet, 900mg , BID
  Arms: Cohort 9
Drug: GS-6620 tablet — GS-6620 tablet, 900 mg
  Arms: Cohort 11

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Multiple Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GS-6620 in Treatment Naïve Subjects with Chronic Hepatitis C Virus Infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-60 years of age or up to 64 years of age with approval)
* Documented chronic HCV infection to be of at least 6 months duration and plasma HCV RNA ≥ 5 log10 IU/mL at screening.
* HCV treatment naïve
* Estimated creatinine clearance ≥ 80 mL/min,
* QTcF interval ≤ 450 msec, QRS duration < 100 msec, PR interval < 220 msec,
* Body mass index (BMI) of 19.0 to 34.0 kg/m2, inclusive.
* Eligible subjects must also be HCV treatment-naïve.

Exclusion Criteria:

* Subjects with prior documentation of cirrhosis, excessive current alcohol intake, any evidence of hepatocellular carcinoma (i.e., α-fetoprotein > 50 ng/mL or by any other standard of care measure)
* Urine drug screen positive for illicit/illegal drugs
* ALT and AST levels > 5 times the upper limit of the normal range (ULN)
* Direct bilirubin > ULN, clinical or other laboratory evidence of hepatic decompensation (i.e., platelets < 100,000/mm3, prothrombin time ≥ 1.5 × ULN and albumin < 3.5 g/dL) are not eligible for study participation.
* Subjects with an absolute neutrophil count (ANC) < 1,000 cells/mm3 (< 750 cells/mm3 for black or African-American subjects), hemoglobin (Hb) < 11 g/dL,
* Coinfected with hepatitis B virus (HBV), human immunodeficiency virus (HIV), or another HCV genotype (other than type 1 for Cohorts 1-5 and type 2 or 3 for Cohort 6) are not eligible for study participation.
* Evidence of hepatocellular carcinoma
* Any sign of decompensated liver disease, including prothrombin time ≥ 1.5 X ULN, platelets < 100,000/mm3 or albumin < 3.5 g/dL at screening OR current or prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy or variceal hemorrhage)
* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* History of a primary gastrointestinal disorder that could interfere with the absorption of the study drug or that could interfere with normal gastrointestinal anatomy or motility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability.
Number of subjects with HCV RNA viral response as a measure of antiviral activity.

SECONDARY OUTCOMES:
Concentrations and pharmacokinetic parameters of GS-6620 and its metabolites will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rossi, PharmD, Study Director — Gilead Sciences
Locations (13):
- United States (12):
  - Advanced Clinical Research Institute, Anaheim, California
  - Axis Clinical Trials, Los Angeles, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Saint Louis University, St Louis, Missouri
  - CRI Worldwide, Philadelphia, Pennsylvania
  - St. Luke Episcopal Hospital, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, LC, Salt Lake City, Utah
  - Charles River Clinical Services Northwest, Tacoma, Washington
- Fundacion De Investigacion De Diego, San Juan, PR, Puerto Rico